CLINICAL TRIAL: NCT02186249
Title: Expanded Access Program With Nivolumab (BMS-936558) in Combination With Ipilimumab (Yervoy®) in Subjects With Unresectable or Metastatic Melanoma
Brief Title: Expanded Access Program With Nivolumab in Combination With Ipilimumab in Patients With Tumors Unable to be Removed by Surgery or Metastatic Melanoma
Acronym: CheckMate218
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-218
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

INTERVENTIONS:
Drug: Nivolumab
Drug: Ipilimumab

SUMMARY:
The purpose of this study is to provide treatment with nivolumab in combination with ipilimumab to subjects who are anti-(CTLA)-4 and anti-PD-1 treatment-naive and have unresectable or metastatic melanoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women 18 years and older
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Histologically-confirmed unresectable stage III or stage IV melanoma, as per American Joint Committee on Cancer (AJCC) staging system, Including mucosal and ocular melanoma
* Subjects must be anti-CTLA-4 treatment-naive and anti-PD-1 treatment-naive. Subjects may have had other prior systemic treatment for localized or metastatic disease
* Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 2 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. There must also be no requirement for high doses of systemic corticosteroids that could result in Immunosuppression (>10 mg/day prednisone equivalent) for at least 2 weeks prior to study drug administration

Exclusion Criteria:

* Active (symptomatic) and not treated brain metastases or leptomeningeal metastases
* Life expectancy < 6 weeks
* Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease
* Subjects who received prior therapy with an anti-CTLA-4, anti-PD-1, anti-PD-L1 or anti-PD-L2, anti-CT137 (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways) or subject is expected to require any other form of systemic antineoplastic therapy while receiving nivolumab

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (57):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - 6501 Truxtun Avenue, Bakersfield, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - 100 UCLA Medical Plaza, Los Angeles, California
  - 514 North Prospect Ave, Redondo Beach, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Angeles Clinic and Research Institute, Santa Monica, California
  - 1325 East Church Street, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Smilow Cancer Hospital at Yale University Cancer Center, New Haven, Connecticut
  - Georgetown-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital, Hollywood, Florida
  - 4500 San Pablo Road South, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - UF Health Cancer Center at Orlando Health, Longwood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - 600 Celebrate Life Parkway, Newnan, Georgia
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Oncology Specialists, SC, Niles, Illinois
  - Local Institution, Louisville, Kentucky
  - Medstar Health Research Institute, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Atlantic Health System, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Tulsa Cancer Institute PLLC, Tulsa, Oklahoma
  - Northwest Cancer Specialists PC, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - St Luke's Hospital, Bethlehem, Pennsylvania
  - Greenville Health System, Easley, South Carolina
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, Midland, Texas
  - Texas Oncology, Paris, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Roanoke, Virginia
  - Shenandoah Oncology Association, Winchester, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Grand River Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - Chuq Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Derived] Hodi FS, Chapman PB, Sznol M, Lao CD, Gonzalez R, Smylie M, Daniels GA, Thompson JA, Kudchadkar R, Sharfman W, Atkins M, Spigel DR, Pavlick A, Monzon J, Kim KB, Ernst S, Khushalani NI, van Dijck W, Lobo M, Hogg D. Safety and efficacy of combination nivolumab plus ipilimumab in patients with advanced melanoma: results from a North American expanded access program (CheckMate 218). Melanoma Res. 2021 Feb 1;31(1):67-75. doi: 10.1097/CMR.0000000000000708. PMID 33234846
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx